CLINICAL TRIAL: NCT03584178
Title: The Long-Term Safety of Budesonide Via Mucosal Atomization Device and Impregnated Nasal Saline Irrigations for Patients With Chronic Rhinosinusitis - A Prospective Double Cohort Study.
Brief Title: The Long-Term Safety of Budesonide for Patients With Chronic Rhinosinusitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Paul's Hospital, Canada (Other)
Responsible Party: Principal Investigator, Amin Javer, Director, St. Paul's Sinus Centre, St. Paul's Hospital, Canada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H18-00458
Record Dates: First submitted 2018-06-18; First posted 2018-07-12 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Sinusitis
Keywords: ACTH-axis; Budesonide; MAD; INSI; Intraocular pressure; Bone density
MeSH Terms: conditions — Sinusitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mucosal Atomization Device (Experimental): Budesonide via MAD Device
  Interventions: Device: Budesonide via MAD device
- Intranasals Saline Irrigation (Experimental): Budesonide via Intranasals Saline Irrigation
  Interventions: Device: Budesonide via intranasals Saline Irrigation

INTERVENTIONS:
Device: Budesonide via MAD device — Delivery through Mucosal Atomization Device
  Other Names: Budesonide via Mucosal Atomization Device
  Arms: Mucosal Atomization Device
Device: Budesonide via intranasals Saline Irrigation — delivery via nasal irrigation bottle
  Other Names: Intranasals Saline Irrigation
  Arms: Intranasals Saline Irrigation

SUMMARY:
Chronic Rhinosinusitis (CRS) is a common disorder of the nose. The current practice at St Paul's Sinus Centre is to prescribe budesonide via the mucosal atomization device or impregnated saline irrigation. Both have shown to be a safe method of administration. A previous study demonstrated a 6% elevation in intraocular pressure and 3% prevalence of asymptomatic AdrenoCorticoTropic Hormone-Axis (ACTH) suppression. However, a baseline measurement was not conducted to ascertain the correlation of these findings with the medication. Therefore, the investigators aim to conduct baseline measurements of IntraOcular Pressure (IOP), ACTH-axis function, and Dual Energy X-ray Absorptiometry (DEXA) scan and obtaining regular measurements of these variables within a 12-month period to further ascertain these previous findings.

DETAILED DESCRIPTION:
Purpose:

The purpose of this study is to assess the long-term effects of budesonide via MAD (Mucosal Atomization Device) or INSI (Intranasal Saline Irrigation) on intraocular pressure, ACTH-axis function, and bone-density.

Hypothesis:

Budesonide delivered via MAD or INSI will be safe in the long-term (> 12 months) demonstrated objectively via IOP, ACTH stimulation test, and DEXA scan.

Justification:

The safety profile of both MAD and INSI has been widely studied in the literature. Although both modalities are generally considered safe, several studies have demonstrated asymptomatic hypothalamic-pituitary-adrenal axis (HPAA) suppression when used in the long-term. A cross-sectional study at St Paul's Sinus Centre, found 3% of study participants on long-term maintenance treatment via MAD to have asymptomatic HPAA suppression. However, the cross-sectional study design limited the ability to ascertain the timeline for this adverse event.

Although the recent cross-sectional study at St Paul Sinus Centre was the first to study the long-term effects of budesonide via the MAD in CRS patients, it did not include baseline levels of HPAA function and IOP levels which served as a limitation to ascertaining the timeline of the aforementioned adverse events. Additionally, there is currently limited data on the effects of INCS on bone function in the setting of CRS treatment. Therefore, this study aims to prospectively assess the long-term effect of high-dose nasal corticosteroids (i.e. INSI and MAD) in CRS patients. The study design will obtain baseline measurements of ACTH function, IOP measurement, and a DEXA scan to identify and describe the timeline of adverse events should they develop during the 12-month study period. By determining the impact of nasal corticosteroids on these outcomes, potential improvements can be made in the safety monitoring practices of otolaryngologists. This may include more frequent monitoring of intraocular pressure, Bone Mineral Density (BMD), and HPAA-axis function in at-risk populations, development of budesonide tapering guidelines, and improved screening of patient-reported adverse events. Overall, the investigators hope the results from this study will be a step forward in the development of screening guidelines for monitoring patients on long-term IntraNasal CorticoSteroids (INCS) therapy.

Primary Objective:

To assess long-term safety (> 12 months) of budesonide delivered via MAD or INSI as measured objectively via IOP, ACTH stimulation test, and DEXA scan.

Research Design:

A Prospective Double-Cohort Study

Statistical Analysis:

Descriptive statistics will be used to analyze the baseline characteristic data and the data from the administered surveys and objective findings of ACTH stimulation test, IOP measurement, and DEXA scans. In addition, rigorous statistical analysis will be conducted on the Likert scale-based SinoNasal Outcome Test (SNOT-22) and EuroQuol health-related quality of life surveys (EQ-5D-5L). These analyses will include cross-tabulations (Pearson's chi square test) and confidence interval calculations. Due to the variations in baseline intraocular pressure measurements, the investigators will calculate an adjusted difference instead of absolute values.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged between 19 years and above
2. Patients with chronic or recurrent sinusitis (as defined by the American Academy of Otolaryngology) with nasal polyposis
3. Patients with an upcoming Functional Endoscopic Sinus Surgery (FESS) procedure
4. Patients being prescribed INCS for the first time following FESS

Exclusion Criteria:

1. Individuals unable to understand the purpose, methods and conduct of this study
2. Patients unwilling to provide informed consent
3. Patients with significant comorbidities (such as tumour, CF, wegeners granulomatosis, immunocompromised)
4. Patients with a history of pituitary disease
5. Patients with a known hypersensitivity to cortisol, corticotropin, or cosyntropin
6. Patients with history of glaucoma or cataracts
7. Recent use of systemic corticosteroids such as prednisone (within last 3 months)
8. Patients that are not adherent to budesonide via MAD/INSI treatment

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-09-05 (Actual); Primary Completion 2020-12-25 (Estimated); Study Completion 2021-12-25 (Estimated)

PRIMARY OUTCOMES:
Sinonasal-Outcomes Test-22 (SNOT-22) Questionnaire | 1 year
  This sinus-specific questionnaire is divided into three parts consisting of 22 questions that are related to sinus health and health-related quality of life. This questionnaire was developed to assess symptoms and quality of life in patients suffering from CRS with or without nasal polyposis. Each question is scored on an ordinal, categorical scale ranging from 0 to 5. Patients are instructed to indicate if symptoms are "absent (0)", "very mild (1)", "mild (2)", "moderate (3)", "severe (4)" or "as bad as it can be (5)". The highest score achievable on this questionnaire is 110 points. Higher scores indicate greater symptom severity and burden on daily life. In a validation survey of 2803 subjects, the SNOT-22 showed high internal consistency, test-retest reliability and validity. The SNOT-22 was found to sufficiently distinguish between patients with CRS and healthy controls (P<0.0001, t=85.3).

CONTACTS AND LOCATIONS:
Overall Officials: Amin Javer, MD, Principal Investigator — University of British Columbia
Locations (1):
- St Paul Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No